CLINICAL TRIAL: NCT02753530
Title: Phase II Study of Arimoclomol for the Treatment of Sporadic Inclusion Body Myositis (IBM)
Brief Title: Study of Arimoclomol in Inclusion Body Myositis (IBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZevraDenmark (Industry)
Collaborators: University of Kansas Medical Center (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002461; R01FD004809 (FDA)
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Inclusion Body Myositis
Keywords: IBM
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — arimoclomol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arimoclomol (Experimental): 248 mg arimoclomol base (equivalent to 400 mg arimoclomol citrate) 3 times daily
  Interventions: Drug: Arimoclomol
- Placebo (Placebo Comparator): 248 mg matching placebo 3 times daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Arimoclomol — 2 capsules (2 x 124 mg arimoclomol base; equivalent to 2 x 200 mg arimoclomol citrate) taken 3 times daily during breakfast, early afternoon, and at bedtime
  Arms: Arimoclomol
Other: Placebo — 2 matched placebo capsules taken 3 times daily during breakfast, early afternoon, and at bedtime
  Arms: Placebo

SUMMARY:
Funding Source - FDA Office of Orphan Products Development (OOPD). The purpose of this study is to evaluate the safety and efficacy of the study drug, arimoclomol in IBM patients.

DETAILED DESCRIPTION:
A Phase 2/3, randomized, double-blind, placebo-controlled, international, 20-month intervention study in patients with IBM.

ELIGIBILITY:
Inclusion Criteria:

* Meet any of the European Neuromuscular Centre Inclusion Body Myositis research diagnostic criteria 2011 categories for IBM.
* Demonstrate being able to arise from a chair without support from another person or device.
* Able to ambulate at least 20 ft/6 meters with or without assistive device. Once arisen from the chair, participant may use any walking device, i.e. walker/frame, can, crutches, or braces. They cannot be supported by another person and cannot use furniture or wall for support.
* Age at onset of weakness >45 years.
* Body weight of >= 40 kg.
* Able to give informed consent.

Exclusion Criteria:

* History of any of the following excludes subject participation in the study: chronic infection particularly HIV or Hepatitis B or C; cancer other than basal cell cancer less than five years prior; or other chronic serious medical illnesses.
* Presence of any of the following on routine blood screening: White blood cells (WBC) <3000; platelets < 100,000; hematocrit <30%; blood urea nitrogen (BUN) >30 mg/dL; creatinine >1.5 x upper limit of normal; symptomatic liver disease with serum albumin <3 g/dL.
* History of most recent creatine kinase >15x the upper limit of normal without any other explanation besides IBM.
* History of non-compliance with other therapies.
* Use of testosterone except for physiologic replacement doses in case of androgen deficiency. Participants must have documented proof of the androgen deficiency.
* Coexistence of other disease that would be likely to affect outcome measures
* Drug or alcohol abuse within past three months.
* Participation in a recent drug study in the last 30 days prior to the screening visit or use of a biologic agent less than 6 months prior to the screening visit.
* Women who are lactating or unwilling to use adequate method of birth control who are not surgically sterile. Adequate birth control includes use of intrauterine device, abstinence, or oral contraceptives or a double barrier method, e.g condom plus diaphragm will be necessary for both male and female participants.
* Participants taking >7.5 mg prednisolone or equivalent or participants on Intravenous Immunoglobulin Therapy (IVIg) or other immunosuppressants within the last 3 months.
* Clinically significant renal or hepatic disease, as indicated by clinical laboratory assessment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, MD, Principal Investigator — University of Kansas Medical Center; Michael Hanna, MD, Principal Investigator — University College, London
Locations (12):
- United States (11):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- University College of London, London, United Kingdom

REFERENCES:
- [Derived] Salam S, Symonds T, Doll H, Rousell S, Randall J, Lloyd-Price L, Hudgens S, Guldberg C, Herbelin L, Barohn RJ, Hanna MG, Dimachkie MM, Machado PM; Members of the Arimoclomol in IBM Investigator Team of the Neuromuscular Study Group. Measurement properties of the Inclusion Body Myositis Functional Rating Scale. J Neurol Neurosurg Psychiatry. 2025 Jan 16;96(2):122-131. doi: 10.1136/jnnp-2024-333617. PMID 38960586
- [Derived] Machado PM, McDermott MP, Blaettler T, Sundgreen C, Amato AA, Ciafaloni E, Freimer M, Gibson SB, Jones SM, Levine TD, Lloyd TE, Mozaffar T, Shaibani AI, Wicklund M, Rosholm A, Carstensen TD, Bonefeld K, Jorgensen AN, Phonekeo K, Heim AJ, Herbelin L, Barohn RJ, Hanna MG, Dimachkie MM; Arimoclomol in IBM Investigator Team of the Neuromuscular Study Group. Safety and efficacy of arimoclomol for inclusion body myositis: a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2023 Oct;22(10):900-911. doi: 10.1016/S1474-4422(23)00275-2. PMID 37739573

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimoclomol (20 Months): Arimoclomol base 248 mg 3 times daily for 20 months
- Placebo (20 Months): Matching placebo 3 times daily for 20 months
Period: Overall Study
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Started | 74 (One patient was randomized in error to arimoclomol but was not treated and was excluded from the intention-to-treat (ITT) and safety populations) | 78 (One patient was randomized in error and was therefore excluded from the intention-to-treat (ITT) population but included in the safety population since exclusion occurred after dosing.)
Completed | 62 | 72
Not Completed | 12 | 6
Not completed — Adverse Event | 7 | 1
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population. Patients randomized in error (1 patient in the arimoclomol group and 1 patient in the placebo group) were not included in the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months) | Total
Number analyzed (Participants) | 73 | 77 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (8.18) | 67.4 (8.08) | 67.2 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 53 | 61 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 72 | 75 | 147
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 69 | 74 | 143
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Age at diagnosis [Mean (Standard Deviation); unit: Years] | 63.4 (8.67) | 63.5 (7.94) | 63.4 (8.28)
Inclusion Body Myositis Functional Rating Scale (IBMFRS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The IBMFRS is a 10-item questionnaire. Scores for each item range from 0 to 4. There is a total maximum score of 40 and minimum score of 0. The higher the score the better functional status of the person.
  score on a scale | 26.88 (4.740) | 27.92 (4.394) | 27.41 (4.581)

OUTCOME MEASURES:

1. Primary Outcome: Change in Inclusion Body Myositis Functional Rating Scale (IBMFRS) Total Score
Description: Measured by rate of decline in the IBMFRS between experimental and placebo groups. The IBMFRS is a 10-item questionnaire. Scores for each item range from 0 to 4. There is a total maximum score of 40 and minimum score of 0. The higher the score the better functional status of the person.
Time Frame: Change from Baseline to Month 20
Population: Intention-to-treat; participants with data at Month 20
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 62 | 72
score on a scale | -3.26 [-4.15 to -2.36] | -2.26 [-3.11 to -1.41]
Statistical Analysis 1: Comparison: Arimoclomol (20 Months) vs Placebo (20 Months); The baseline observation was the last observation recorded prior to the first dose of study medication. The change from baseline in IBMFRS total score was analyzed using a Mixed Models for Repeated Measures (MMRM) with treatment interacting with visit and trial site as factors. Baseline IBMFRS total score interacting with visit was further included as covariate. An unstructured covariance matrix was assumed; Test type: Superiority; p = 0.1146, Mixed Models Analysis — Primary Estimand (Treatment Policy); Least Square (LS) Mean Difference = -0.99, 95% CI 2-sided [-2.23 to 0.24]

2. Secondary Outcome: Change in Inclusion Body Myositis Functional Rating Scale (IBMFRS) Total Score
Description: as for outcome 1
Time Frame: Change from Baseline to Month 12
Population: Intention-to-treat; participants with data at Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 63 | 73
score on a scale | -1.87 (3.494) | -1.03 (3.127)

3. Secondary Outcome: Grip Strength
Description: Unilateral hand grip strength in both hands measured using the Jamar Dynamometer. Results are for the stronger limb, as identified at baseline.
Time Frame: Change from Baseline to Month 12 and 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
kg
  Change from Baseline to Month 12: number analyzed (Participants) | 58 | 67
  Change from Baseline to Month 12 | -1.09 (5.459) | -1.84 (3.259)
  Change from Baseline to Month 20: number analyzed (Participants) | 56 | 68
  Change from Baseline to Month 20 | -3.93 (9.201) | -2.86 (4.741)

4. Secondary Outcome: Modified Timed up and go (mTUG)
Description: The patient's combined ability to rise from a chair and walk 3 meters, turn around and walk back to the chair and sit down. The test was performed twice and the fastest time was used. The results were expressed as velocity in meters/second.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: meters per second (m/sec)
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
meters per second (m/sec)
  Change from Baseline to Month 12: number analyzed (Participants) | 60 | 67
  Change from Baseline to Month 12 | -0.075 (0.3048) | -0.058 (0.2281)
  Change from Baseline to Month 20: number analyzed (Participants) | 57 | 67
  Change from Baseline to Month 20 | -0.084 (0.1893) | -0.104 (0.1955)

5. Secondary Outcome: Manual Muscle Testing (MMT), Total Score
Description: The Manual Muscle Testing (MMT) scores the strength of 24 muscles (axial, proximal, and distal muscles, tested bilaterally) on a scale from 0 to 10 points. The total score is calculated as an average across the 24 muscles and ranges from 0 to 10. The total score will increase if a patient is getting stronger and decrease if a patient is getting weaker.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
score on a scale
  Change from Baseline to Month 12: number analyzed (Participants) | 60 | 67
  Change from Baseline to Month 12 | -0.49 (0.878) | -0.47 (0.855)
  Change from Baseline to Month 20: number analyzed (Participants) | 57 | 68
  Change from Baseline to Month 20 | -0.48 (0.922) | -0.53 (0.764)

6. Secondary Outcome: 6 Minute Walk Test (6MWT); Distance After 6 Minutes (6MWD)
Description: The distance patients could walk in 6 minutes. The distance walked in meters was recorded after 6 minutes.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
meters
  Change from Baseline to Month 12: number analyzed (Participants) | 56 | 65
  Change from Baseline to Month 12 | -16.7 (56.24) | -10.7 (43.65)
  Change from Baseline to Month 20: number analyzed (Participants) | 52 | 66
  Change from Baseline to Month 20 | -37.0 (80.09) | -30.9 (65.68)

7. Secondary Outcome: Short Form-36 (SF-36) Physical Component Score
Description: Measured using the Short Form health survey with 36 items (SF-36). The questionnaire measures 8 health concepts which yields 2 summary measures: physical and mental health. The physical component score includes 4 scales of physical functioning (10 items), role limitations due to physical health (4 items), bodily pain (2 items), and general health (5 items). To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100, and the summary measure is calculated as the average score. Higher scores indicate better health status.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: score on a scale (physical component)
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
score on a scale (physical component)
  Change from Baseline to Month 12: number analyzed (Participants) | 61 | 71
  Change from Baseline to Month 12 | -1.3 (5.39) | -2.0 (6.21)
  Change from Baseline to Month 20: number analyzed (Participants) | 61 | 69
  Change from Baseline to Month 20 | -1.0 (6.94) | -3.4 (6.51)

8. Secondary Outcome: Maximum Voluntary Isometric Contraction (MVICT) of Quadriceps
Description: Unilateral strength of the knee extensor muscles on both limbs using the MicroFET hand-held dynamometer. Results are for the stronger limb, as identified at baseline.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
kg
  Change from Baseline to Month 12: number analyzed (Participants) | 57 | 66
  Change from Baseline to Month 12 | -2.59 (9.357) | -2.49 (6.067)
  Change from Baseline to Month 20: number analyzed (Participants) | 55 | 67
  Change from Baseline to Month 20 | -6.29 (12.013) | -4.67 (7.885)

9. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: The disability index of the HAQ measures self-reported functional status (disability) including the patient's use of aids or devices and/or help from other persons. The scale is composed of 20 items in 8 domains (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities). Each domain has at least 2 subcategory items, scored on a scale from 0 to 3, and for each of the 8 domains the domain score was the highest score of the involved subcategory scores. The total score reported is an average over 8 domains and scores from at least 6 domains had to be available for the total score to be calculated. The average total score ranges from 0 to 3, and a higher score corresponds to a worsening in functional status.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
score on a scale
  Change from Baseline to Month 12: number analyzed (Participants) | 63 | 73
  Change from Baseline to Month 12 | 0.24 (0.364) | 0.24 (0.375)
  Change from Baseline to Month 20: number analyzed (Participants) | 60 | 70
  Change from Baseline to Month 20 | 0.33 (0.399) | 0.33 (0.472)

10. Secondary Outcome: 2 Minute Walk Test (2MWT)
Description: The distance patients could walk in 2 minutes (during the 6 Minute Walk Test) recorded in meters.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
meters
  Change from Baseline to Month 12: number analyzed (Participants) | 54 | 64
  Change from Baseline to Month 12 | -4.73 (19.355) | -2.40 (16.789)
  Change from Baseline to Month 20: number analyzed (Participants) | 51 | 66
  Change from Baseline to Month 20 | -11.18 (25.551) | -8.52 (23.601)

11. Secondary Outcome: Short Form-36 (SF-36) Mental Component Score
Description: Measured using the Short Form health survey with 36 items (SF-36). The questionnaire measures 8 health concepts which yields 2 summary measures: physical and mental health. The mental component score is composed of energy/fatigue (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and emotional well-being (5 items). To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100, and the summary measure is calculated as the average score. Higher scores indicate better health status.
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Mean (Standard Deviation); unit: score on a scale (mental component)
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
score on a scale (mental component)
  Change from Baseline to Month 12: number analyzed (Participants) | 61 | 71
  Change from Baseline to Month 12 | -2.0 (7.00) | -2.1 (7.47)
  Change from Baseline to Month 20: number analyzed (Participants) | 61 | 69
  Change from Baseline to Month 20 | -2.5 (9.19) | -1.3 (7.08)

12. Secondary Outcome: Patient Global Impression of Severity (PGIS)
Description: Patient-reported assessment of the impact of IBM on the ability to complete activities of daily living (e.g. dressing, walking, bathing) at the time of the assessment. The response options for the impact of IBM were "none" (i.e. no impact), "very mild", "mild", "moderate", "severe", and "very severe".
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 56 | 66
Participants
  Month 12: None | 0 | 1
  Month 12: Very mild | 1 | 3
  Month 12: Mild | 9 | 12
  Month 12: Moderate | 31 | 40
  Month 12: Severe | 14 | 10
  Month 12: Very severe | 1 | 0
  Month 20: None | 0 | 1
  Month 20: Very mild | 2 | 2
  Month 20: Mild | 8 | 8
  Month 20: Moderate | 26 | 43
  Month 20: Severe | 19 | 12
  Month 20: Very severe | 1 | 0

13. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient-reported assessment of the change from start of study treatment in the impact of IBM on the ability to complete activities of daily living (e.g. dressing, walking, bathing). The response options for change in impact were "very much worse", "much worse", "a little worse", "no change", "a little improved", "much improved", and "very much improved".
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 56 | 66
Participants
  Month 12: Very much worse | 1 | 0
  Month 12: Much worse | 10 | 8
  Month 12: A little worse | 27 | 43
  Month 12: No change | 12 | 13
  Month 12: A little improved | 4 | 1
  Month 12: Much improved | 2 | 0
  Month 12: Very much improved | 0 | 0
  Month 12: Missing | 0 | 1
  Month 20: Very much worse | 4 | 2
  Month 20: Much worse | 23 | 16
  Month 20: A little worse | 19 | 40
  Month 20: No change | 5 | 6
  Month 20: A little improved | 3 | 2
  Month 20: Much improved | 2 | 0
  Month 20: Very much improved | 0 | 0
  Month 20: Missing | 0 | 0

14. Secondary Outcome: Clinician Global Impression of Severity (CGIS)
Description: Clinician-reported assessment of the severity of the patient's IBM symptoms at the time of the assessment. The response options were "none", "very mild", "mild", "moderate", "severe", and "very severe"
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 5 | 9
Participants
  Month 12: None | 0 | 0
  Month 12: Very mild | 0 | 0
  Month 12: Mild | 0 | 2
  Month 12: Moderate | 2 | 4
  Month 12: Severe | 1 | 0
  Month 12: Very severe | 0 | 0
  Month 12: Missing | 2 | 3
  Month 20: None | 0 | 0
  Month 20: Very mild | 1 | 0
  Month 20: Mild | 1 | 2
  Month 20: Moderate | 2 | 2
  Month 20: Severe | 1 | 3
  Month 20: Very severe | 0 | 0
  Month 20: Missing | 0 | 2

15. Secondary Outcome: Clinician Global Impression of Change (CGIC)
Description: Clinician-reported assessment of the change from start of study treatment in the patient's IBM symptoms. The response options for change in IBM were "very much worse", "much worse", "a little worse", "no change", "a little improved", "much improved", and "very much improved".
Time Frame: Change from Baseline to Month 12 and Month 20
Population: Intention-to-treat; participants with data at Month 12 and Month 20, respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 5 | 9
Participants
  Month 12: Very much worse | 0 | 0
  Month 12: Much worse | 1 | 0
  Month 12: A little worse | 2 | 5
  Month 12: No change | 0 | 0
  Month 12: A little improved | 0 | 1
  Month 12: Much improved | 0 | 0
  Month 12: Very much improved | 0 | 0
  Month 12: Missing | 2 | 3
  Month 20: Very much worse | 0 | 0
  Month 20: Much worse | 0 | 1
  Month 20: A little worse | 3 | 4
  Month 20: No change | 2 | 0
  Month 20: A little improved | 0 | 1
  Month 20: Much improved | 0 | 1
  Month 20: Very much improved | 0 | 0
  Month 20: Missing | 0 | 2

16. Secondary Outcome: Falls and Near Falls
Description: Falls and near falls registered by the participants in a diary
Time Frame: Accumulated number from Baseline to Month 20
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: events (falls or near-falls) per year
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
Number analyzed (Participants) | 73 | 77
events (falls or near-falls) per year
  Falls/year | 4.8 (5.43) | 5.8 (11.71)
  Near-falls/year | 9.1 (28.52) | 6.9 (17.12)

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 14 days following the latest administration of study medication. Assessed monthly for the first 6 months, and then every second month until Month 20.
Description: The safety population included all participants who received any amount of study medication.
  The safety analysis included all events occurring during the on-treatment observation period which started at the date of first administration of study medication and until 14 days following the latest administration of study medication. The results are similar to those during the in-trial period (from written informed consent until the telephone follow-up visit, 30 days after the end of the trial).
Arm/Group | Arimoclomol (20 Months) | Placebo (20 Months)
All-Cause Mortality (participants affected / at risk) | 1/73 | 1/78
Serious Adverse Events (participants affected / at risk) | 11/73 | 18/78
Other Adverse Events (participants affected / at risk) | 72/73 | 70/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (20 Months) (N=73) | Placebo (20 Months) (N=78)
Bursitis infective (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chronic hepatitis B (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (20 Months) (N=73) | Placebo (20 Months) (N=78)
Contusion (Injury, poisoning and procedural complications) | 8 | 13
Fall (Injury, poisoning and procedural complications) | 7 | 6
Laceration (Injury, poisoning and procedural complications) | 6 | 8
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 5 | 7
Foot fracture (Injury, poisoning and procedural complications) | 4 | 6
Joint injury (Injury, poisoning and procedural complications) | 2 | 7
Limb injury (Injury, poisoning and procedural complications) | 2 | 4
Rib fracture (Injury, poisoning and procedural complications) | 0 | 4
Nasopharyngitis (Infections and infestations) | 10 | 13
Upper respiratory tract infection (Infections and infestations) | 6 | 11
Sinusitis (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 2 | 5
Influenza (Infections and infestations) | 4 | 2
Constipation (Gastrointestinal disorders) | 14 | 9
Diarrhoea (Gastrointestinal disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 9 | 1
Dry mouth (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Blood creatinine increased (Investigations) | 9 | 1
Weight decreased (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 6 | 3
Headache (Nervous system disorders) | 7 | 4
Dizziness (Nervous system disorders) | 8 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 1
Paraesthesia (Nervous system disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 4
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0
Fatigue (General disorders) | 8 | 3
Oedema peripheral (General disorders) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Gout (Metabolism and nutrition disorders) | 0 | 4
Alcohol intolerance (Metabolism and nutrition disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hypertension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02753530/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT02753530/SAP_001.pdf